CLINICAL TRIAL: NCT01862627
Title: Macular Retinoschisis and Detachment Associated With Glaucomatous Optic Neuropathy But Without Optic Disc Pit Nor High Myopia
Brief Title: Macular Retinoschisis and Detachment Associated With Glaucomatous Optic Neuropathy
Status: Completed | Type: Observational
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Associate professor of ophthalmology, Kyorin University
Other Study IDs: Kyorineye011
Record Dates: First submitted 2013-05-15; First posted 2013-05-24 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Macular Retinoschisis; Macular Detachment; Normal Tension Glaucoma
Keywords: Macular retinoschisis; Macular detachment; vitrectomy
MeSH Terms: conditions — Low Tension Glaucoma | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Macular retinoschisis and detachment
  Interventions: Procedure: Optical coherence tomography

INTERVENTIONS:
Procedure: Optical coherence tomography

SUMMARY:
Clinical features, optical coherence tomography findings and surgical outcome in eyes with macular retinoschisis and detachment with normal tension glaucoma but without optic disc pit or high myopia were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The patients with macular retinoschisis and detachment associated with normal tension glaucoma

Exclusion Criteria:

* Optic pit maculopathy, high myopia

Ages: 10 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients with macular retinoschisis and detachment associated with normal tension glaucoma
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2004-12; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Optical coherence tomography | One year
  Anatomical improvement detected with optical coherence tomography after surgical intervention.

SECONDARY OUTCOMES:
Visual recovery | One year
  The number of the patients with visual recovery after surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Inoue, MD, Principal Investigator — Kyorin Eye Center
Locations (1):
- Kyorin Eye Center, Mitaka, Tokyo, Japan